CLINICAL TRIAL: NCT04370912
Title: Using Bedside Ultrasound to Screen for Sarcopenia in Older Adults
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Kenneth Madden, Allan M. McGavin Chair in Geriatric Medicine Division Head, Vancouver General Hospital Division of Geriatric Medicine, University of British Columbia
Other Study IDs: H20-01355
Record Dates: First submitted 2020-04-27; First posted 2020-05-01 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Hand Strength

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bed side Ultrasound — Handgrip strength will be measured using a digital grip strength dynamometer (Sammons Preston, Nottinghamshire, UK). This measurement is carried out three times using the subject's dominant hand, and then averaged
  Other Names: Grip strength; Appendicular Skeletal Mass assessment

SUMMARY:
The loss of both muscle mass and quality with increasing age is called 'sarcopenia' and is a risk factor for falls, fractures and increased mortality. Sarcopenia is diagnosed with Dual-energy X-ray absorptiometry (DXA) scanning (according to current criteria), but in Canada DXA scans are not approved to screen for this condition. One potential solution is Point of Care Ultrasound (PoCUS), since recent advances have made bedside ultrasound technology readily available as a rapid bedside screening tool.

DETAILED DESCRIPTION:
Some recent work has examined the possibility of using ultrasound as a measure of both muscle quantity and muscle quantity. Work done by Strasser et al, has shown that ultrasonic measures of muscle thickness in the quadriceps muscle has a highly significant correlation with maximal voluntary contration. Other work done by Miron-Mombiela et al has shown that measures of muscle thickness and echointensity (a measure of muscle quality) also show high correlations with grip strength. These findings (supported by our pilot data, see Pilot Data) and new technological advances in bedside ultrasonic devices suggest that these measures might be a valuable contribution to the process of screening for sarcopenia in older adults. In this proposal, Investigators hypothesize that bedside ultrasound, which is increasingly becoming a mainstream component of the standard physical exam, will be a much more specific and accurate alternative to our current best screening methods.

ELIGIBILITY:
Inclusion Criteria:

* each subject must be 65 years of age or greater

Exclusion Criteria:

* hemodialysis patients will be excluded, due to excessive fluid shifts with dialysis
* patients using chronic oral corticosteroids will be excluded, due to potential muscle atrophy
* hemiparesis due to a stroke or paresis of the lower limbs will be excluded
* subjects with pitting edema on physical exam (due to liver, renal or heart failure) or patients that are severely dehydrated will be excluded
* patients with myositis, systemic connective tissue disorders, systemic atrophies affecting the central nervous system (CNS) and CNS demyelinating diseases will be excluded

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Subjects will be recruited from Vancouver Coastal Health Authority has 5 outpatient geriatric medicine clinics that continuously for 5 days per week and see 4000 new patients per year.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
US measurement for Sarcopenia | through study completion, an average of 1 year
  o establish PoCUS measures (muscle thickness, MT; echointensity, EI) as a new screening test for sarcopenia
Weight in kg | through study completion, an average of 1 year
  weight and height will be combined to report BMI in kg/m^2
Height in cm | through study completion, an average of 1 year
  weight and height will be combined to report BMI in kg/m^2
Handgrip strength in kg | through study completion, an average of 1 year
  Handgrip strength cutoffs for sarcopenia for men and women

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Madden, MD, Principal Investigator — UBC
Locations (1):
- Vancouver Coastal Health Research Institute, VGH Research Pavilion Room 186, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided